CLINICAL TRIAL: NCT05162638
Title: Analysis of Lymphatic Fluid From the Thoracic Duct of Healthy People and People With Multiple Sclerosis (MS) Before and After Ofatumumab Treatment
Brief Title: Immune Profiles in Multiple Sclerosis (MS) Patients and Healthy Volunteers Through Thoracic Duct Cannulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Novartis Institutes for BioMedical Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 849114
Record Dates: First submitted 2021-11-02; First posted 2021-12-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; Healthy
Keywords: multiple sclerosis; thoracic duct
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 'In-and-out' catheterization (Other): Safety and immune-cell profile of lymphatic fluid in MS patients with a single time-point sampling of lymphatic fluids and peripheral blood compared to healthy controls.
  Two healthy controls and six patients with early MS (never treated or at least 90 days after discontinued treatment with glatiramer acetate or interferons), who consent to the 'In-and-out' catheter procedure. MS participants can also consent to OMB treatment with 2-year follow-up.
  Interventions: Procedure: thoracic duct cannulation
- "Indwelling" catheterization (Other): immune-biology in people with MS before and during/after OMB treatment within thoracic duct and peripheral blood via indwelling catheter and multiple time-point sampling compared to healthy controls (without drug treatment).
  Twelve patients with early MS (never treated or at least 90 days after discontinued treatment with glatiramer acetate or interferons), who consent to treatment with OMB and to the indwelling catheter procedure with serial sampling and up to four healthy controls (no drug treatment)
  Interventions: Procedure: thoracic duct cannulation

INTERVENTIONS:
Procedure: thoracic duct cannulation — Contrast is injected into lymph nodes until lymphatics visualized at about level of L3 lumbar spine. After target lymphatic vessel is identified, needle is passed transabdominally into the vessel. Guidewire is advanced through the needle into the lymph vessel & advanced into thoracic duct. Microcatheter is then advanced into thoracic duct over the wire.
  IN & OUT-up to 100mL collected via catheter over 30-min at 2 levels within thoracic duct, then catheter removed.
  INDWELLING-As described above, then guidewire placed through original catheter & advanced into subclavian vein. Vascular sheath is placed into vein in the upper arm under ultrasound/fluoroscopy guidance. Wire in the subclavian vein then snared through venous access sheath & pulled out. Catheter then threaded & advanced over the wire until tip is in thoracic duct. Catheter from thoracic duct removed, leaving catheter extending from arm into thoracic duct. Catheter left in place up to 21 days for sampling.

SUMMARY:
In this study, lymph fluid will be collected by cannulation of the thoracic duct, a minimally invasive procedure performed by interventional radiologists. Single time point and serial collection through an indwelling cannula will allow for comparisons between immune cells in the periphery and deep lymphatic system in MS and healthy controls and in MS, changes in responses to a FDA approved therapy ofatumumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for inclusion in this study must meet all of the following criteria:

  1. Written informed consent must be obtained before any assessment is performed.
  2. Adult participants aged 18 to 40 years (inclusive) at Screening.
  3. Participants must be able to understand English and be able to review and comprehend the informed consent form independently or with the help of research staff
  4. No use of systemic glucocorticoids in the past 4 weeks

For participants with MS following additional criteria need to be met:

1. Diagnosis of MS according to the 2017 Revised McDonald criteria.
2. Ability to undergo several MRIs
3. Disability status at Screening with an EDSS score of 0 to 4 (inclusive)
4. MS treatment history restricted to Interferons and/glatiramer acetate treatment only or untreated to date
5. Neurologically stable within one month prior to interventional procedure.

Exclusion Criteria:

* 1. Participants suspected of not being able or willing to cooperate or comply with study protocol requirements in the opinion of the investigator.

  2. Participants with primary progressive MS (Polman C et al., 2011) 3. Participants meeting criteria for neuromyelitis optica (Wingerchuck D et al., 2015) 4. Participants with disease duration of more than 10 years 5. Participants who are pregnant or nursing (lactating) 6. Participants with active chronic disease (or stable but treated with immune therapy) of the immune system other than MS (e.g. rheumatoid arthritis, scleroderma, Sjögren's syndrome, Crohn's disease, ulcerative colitis, etc.) or with immunodeficiency syndrome (hereditary immune deficiency, drug-induced immune deficiency) 7. Participants with active systemic bacterial, viral or fungal infections, or known to have acquired immunodeficiency syndrome (AIDS) 8. Participants with neurological symptoms consistent with PML or confirmed PML 9. Participants at risk of developing or having reactivation of syphilis or tuberculosis 10. History of cardiovascular disease or uncontrolled hypertension 11. History of diabetes mellitus 12. History of cancer (other than localized skin cancer) in the previous 5 years 13. Have received any live or live-attenuated vaccines (including for varicella-zoster virus or measles) within 2 months prior to first study drug administration 14. Immunization with non-live vaccines within 2 weeks of the study procedure 15. Participants at risk of developing or having reactivation of hepatitis: Positive results at Screening for serological markers for hepatitis (H) B and C indicating acute or chronic infection:
  1. HBs Ag and/or anti-HBc IgM and/or HB virus deoxyribonucleic acid (DNA)
  2. anti-HBs negative and Anti-HBc positive
  3. anti-HC IgG (if positive IgG, HCV-RNA PCR will be performed and if negative, participant can be enrolled) 16. Use of other investigational drugs at the time of enrollment (Screening) or within the prior 30 days, or five elimination half-lives, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer 17. Absolute neutrophil count (ANC) <750/mm3; 18. Hemoglobin <10.0 g/dL 19. Platelet count <100,000/mm3 20. Prothrombin time (PT) or international normalized ration (INR) >1.5 x ULN

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | up to 21 days
  Quantified as percent of the study population experiencing serious adverse event from in-and-out catherization procedure and from "indwelling" catheterization procedure
B Cells | up to 21 days
  Change in proportion of flow cytometry defined naïve (CD27-) and memory (CD27+) B cells in thoracic duct of patients with MS prior to and following anti-CD20 therapy with Ofatumumab

SECONDARY OUTCOMES:
Immune cell profiles (MS and healthy controls) | up to 21 days
  Comparison of immune cell profiles determined by flow cytometry of lymphatic fluid and blood between MS and healthy controls
Immune cell profiles (ofatumumab) | up to 21 days
  Comparison of immune cell profiles determined by flow cytometry of lymphatic fluid and blood of MS patients prior to and following treatment with the anti-CD20 Ofatumumab

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bar-Or, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT05162638/Prot_SAP_000.pdf